CLINICAL TRIAL: NCT01756768
Title: A Phase One Open-Label Single-Radiolabeled Dose Study To Investigate The Absorption, Metabolism, And Excretion Of [14C] PD-0332991 In Healthy Male Volunteers
Brief Title: A Single-Radiolabeled Dose Mass Balance Study To Investigate The Absorption, Metabolism, And Excretion Of [14C] Palbociclib (PD-0332991) In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5481011
Record Dates: First submitted 2012-12-20; First posted 2012-12-27 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Phase 1; Mass Balance study; Radio-labeled dose; PD-0332991

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radio-labeled Dose Arm (Experimental)
  Interventions: Radiation: [14C]-PD-0332991

INTERVENTIONS:
Radiation: [14C]-PD-0332991 — A single 125 mg oral dose of PD-0332991 containing approximately 100 microcurie of [14C]-PD-0332991.

SUMMARY:
This will be an open-label, single-center study to evaluate the mass-balance and pharmacokinetics of PD-0332991 in approximately 6 healthy male subjects receiving a single oral 125 mg dose of PD-0332991 containing approximately 100 microcuries of [14C]-PD-0332991. Subjects will be checked in to the research unit from approximately 12 hours prior to dosing and remain in house until greater than 90% of the administered radioactivity is collected from bodily excreta or until less than 1% of the administered radioactivity is recovered from excreta on consecutive days. This study will investigate the extent of involvement of the renal and hepatic systems in the elimination of PD-0332991 and will seek to identify the compound's major metabolites.

ELIGIBILITY:
Inclusion Criteria:

* A Healthy Male Volunteer between 18 and 55 years of age inclusive
* A Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight >50kg
* A signed informed consent document

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular,hepatic,psychiatric, neurologic, or allergic disease.
* A positive urine drug or urine cotinine screen.
* Concurrent use of herbal or prescription medications or treatment with an investigational drug within 30 days or 5 half-lives preceding first dose of study medication.
* Subjects whose occupation requires exposure to radiation or monitoring of radiation exposure.
* Subjects with a history of irregular bowel movements (eg, regular episodes of diarrhea or constipation, irritable bowel syndrome (IBS) or lactose intolerance).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] of PD-0332991 | 0-192 hrs
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PD-0332991 | 0-192hrs
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) of PD-0332991 | 1-24hrs
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PD-0332991 | 1-24hrs
Plasma Decay Half-Life (t1/2) of PD-0332991 | 0-192hrs
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) of PD-0332991 | 0-192hrs
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) of PD-0332991 | 0-192hrs
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Cumulative radioactivity recovery in urine. | 0-192hrs
  Cumulative radioactivity recovered in urine is the percent of the administered radioactive dose that is observed in the cumulative urine samples.
Cumulative radioactivity recovery in feces. | 0-192hrs
  Cumulative radioactivity recovered in fecal is the percent of the administered radioactive dose that is observed in the cumulative fecal samples.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] of PF-05089326. | 0-192hrs
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-05089326. | 0-192hrs
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Plasma Concentration (Cmax) of PF-05089326. | 0-192hrs
Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-05089326. | 0-192hrs
Plasma Decay Half-Life (t1/2) of PF-05089326. | 0-192hrs
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] of radioactivity in plasma. | 0-192hrs
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of radioactivity in plasma. | 0-192hrs
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Maximum Observed Concentration (Cmax) of radioactivity in plasma. | 0-192hrs
Time to Reach Maximum Observed Concentration (Tmax) of radioactivity in plasma. | 0-192hrs
Plasma Decay Half-Life (t1/2) of radioactivity in plasma. | 0-192hrs
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Oral Clearance (CL/F) of radioactivity in plasma. | 0-192hrs
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) of radioactivity in plasma. | 0-192 hrs
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tacoma, Washington, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481011&StudyName=A%20Single-Radiolabeled%20Dose%20Mass%20Balance%20Study%20To%20Investigate%20The%20Absorption%2C%20Metabolism%2C%20And%20Excretion%20Of%20%5B14C%5D%20Palbociclib%20%28PD-0332